CLINICAL TRIAL: NCT03603535
Title: Prospective Study of the sensiTVT (Midurethral Sling) for the Surgical Treatment of Stress Urinary Incontinence
Brief Title: Prospective Study of the sensiTVT
Acronym: sensiTVT
Status: Terminated | Type: Observational
Why Stopped: The recruitment proceeded much slower than expected. The planned number of patients could not be reached within the planned time.
Sponsor: Medical University of Graz (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 29-481 ex 16/17
Record Dates: First submitted 2018-07-05; First posted 2018-07-27 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress urinary incontinence; objective outcome
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: sensiTVT — The study is designed as a prospective single arm study. All women with an indication for suburethral tape placement for therapy of SUI and meeting the inclusion criteria will be offered study participation to record the objective outcome after one year.

SUMMARY:
sensiTVT is a relatively new tape. The aim of this study is to analyze the objective and subjective outcome at one year follow-up.

DETAILED DESCRIPTION:
Stress urinary incontinence (SUI) is defined as the involuntary leakage during physical activity and situations that result in an increase of abdominal pressure like sneezing, coughing or laughing and affects up to 25% of women. Currently there are a number of tapes on the market with GYNECARE TVT EXACT® (Tension free Vaginal Tape) and TVT- Obturator being one of the tapes with the highest subjective and objective cure rates and relatively low adverse events in women with normal sphincter pressure. Due to the recent FDA announcements several tapes have been withdrawn from the market and several new ones have been designed. Data from other tapes are available, however data especially from newer tapes is lacking.

ELIGIBILITY:
Inclusion criteria

* Planned surgery for verified predominant stress urinary incontinence
* women between 18 and 80 years of age
* good German language skills
* informed consent

Exclusion criteria:

* Pregnant or lactating women
* Active surgical treatment for invasive malignant diseases within 3 months
* Contraindications for surgery or anesthesia
* Severe neurologic disease
* Concomitant prolapse surgery

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women with stress urinary incontinence (SUI)
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
objective success of stress urinary incontinence | one year
  determined by a standardized cough stress test at 300 ml bladder, a negative cough stress test is a success.

SECONDARY OUTCOMES:
Subjective success as determined using the Patient Global Impression of Improvement questionnaire. | 3 months+ one year
  defined as very much improved/much improved (1,2) on the Patient Global Impression of Improvement scale, while any other response (improved, same, worse, or much worse- 3-7) will be considered as failures.
  The Patient Global Impression of Improvement is a seven item scale validated for incontinence.
Peri- and postoperative complications | 3 months+ one year
  any surgical complications recorded
Subjective incontinence cure rate using the Incontinence Outcome Questionnaire | 3 months+ one year
  The Incontinence Outcome Questionnaire was validated for postoperative assessment of quality of life after surgical treatment for stress urinary incontinence and has 27 items with lower scores indicating worse treatment outcome. The total score is calculated.
quality of life using the Kings Health Questionnaire | 3 months+ one year
  The Kings Health Questionnaire was validated in women with stress urinary incontinence and assesses the impact of incontinence on quality of life. The eight subscales ("domains") scored between 0 (best) and 100 (worst). The Symptom Severity scale is scored from 0 (best) to 30 (worst); lower scores indicate better QoL. Success in terms of the study is defined as 10 points improvement on the total Kings Health Questionnaire score.
Subjective bother using the Patient Global Impression of Severity | 3 months+ one year
  Patient Global Impression of Severity The Patient Global Impression of Severity is a 7-item urinary symptom severity scale that is used to rate the severity of a specific condition -a single-state scale. The higher the number the worse the outcome of subjective bother of stress urinary incontinence.
Patient satisfaction measured using a visual analogue scale | 3 months+ one year
  Patient satisfaction is defined as a score 8 to 10 on a 10-point visual analogue scale
Sexual health using the Pelvic Organ Prolapse Incontinence Sexual Questionnaire | 3 months+ one year
  The Pelvic Organ Prolapse Incontinence Sexual Questionnaire is a 20 item questionnaire and is the primary measure used to assess sexual function in women with urinary incontinence and prolapse. Mean subscale scores are calculated by summing the valid responses to items in the subscale and then divided by the number of items with valid responses. The higher the subscores, the worse the outcome.
Erosion rate | 3 months+ one year
  Erosion rate from the tape in the vagina or bladder
Reoperation rate | 3 months+ one year
  Reoperation rate
De novo urgency | 3 months+ one year
  De novo OAB- overactive bladder as determined by clinical history taking
De novo pain in the operated region | 3 months+ one year
  De novo pain in the operated region as determined by clinical history taking

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Gold (prev. Ulrich), MD PhD, Principal Investigator — Universitätsklinik für Frauenheilkunde und Geburtshilfe
Locations (1):
- Department of Obstetrics, Medical University Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No